CLINICAL TRIAL: NCT03438565
Title: Safety and Utility Profile of the Asahi Chikai Black 18 neuRovascular guidewirE in Large Vessel Occlusive Stroke: SURE 18 Registry
Brief Title: SURE 18 Registry -Asahi Chikai Black 18 in LVO Stroke
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Asahi Intecc USA Inc (Industry)
Responsible Party: Principal Investigator, Reade A De Leacy, Assistant Professor of Neurosurgery and Radiology; Director of Neurointerventional Spine, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 17-2723
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Occlusive Stroke
Keywords: Asahi Chikai Black 18 Neurovascular Guidewire; Prospective; Retrospective

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Participants with intracranial large vessel occlusive stroke: 50 patients who have been treated with the Asahi Chikai Black 18 neurovascular guidewire.
  Interventions: Device: Asahi Chikai Black 18 neurovascular guidewire
- Historical Control Group: The historical control will include 50 retrospective consecutive patients (who fulfill inclusion and exclusion criteria) treated for acute anterior circulation large vessel occlusive stroke prior to the initiation of the Sure -18 registry.

INTERVENTIONS:
Device: Asahi Chikai Black 18 neurovascular guidewire — The Asahi Chikai Black 18 microguidewire employs a reverse tapered shaft with 0.018" tip and 0.014" proximal shaft, which provides additional support and tactile feedback.
  Groups: Participants with intracranial large vessel occlusive stroke

SUMMARY:
The objective of this study is to obtain post market data on the Asahi Chikai Black 18 neurovascular guidewire in the treatment of intracranial large vessel occlusive stroke. This will be compared to a historical control that will include the prior 50 consecutive patients fitting the same selection criteria.

DETAILED DESCRIPTION:
This is a prospective registry collecting information on 50 patients treated with the ASAHI Chikai Black 18 microguidewire. Patients will undergo mechanical thrombectomy for acute large vessel occlusive stroke within the anterior circulation as is standard of care.

Additionally, this study will have a retrospective portion which will examine 50 consecutive patients who meet inclusion/exclusion criteria treated for acute anterior circulation large vessel occlusive stroke prior to the initiation of the Sure -18 Registry. This retrospective cohort will be 50 consecutive mechanical thrombectomy cases performed using any neurovascular microguidewire other than the device under study (Asahi Chikai Black 18) at the same enrolling centers leading up to December 10, 2018.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients presenting with acute anterior cerebral circulation large vessel occlusive stroke
* ASPECT score 5 or better
* Occlusion of the ICA terminus and M1 MCA
* Favorable CT perfusion with clinical/radiologic mismatch
* Last known well out to 24 hours
* Age limit >18 years
* Baseline mRS 0-3

Exclusion Criteria:

* Intracranial hemorrhage
* ASPECTS (Alberta stroke program early CT score) <5
* Unfavorable CT perfusion
* Baseline mRS 4 or greater
* Large vessel occlusive stroke with tandem lesion of the cervical internal carotid artery or posterior circulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the prospective portion, patients will be enrolled if their doctor decides to treat them with the ASAHI Chikai Black 18 Neurovascular Guidewire.
  For the retrospective portion, 50 consecutive mechanical thrombectomy cases will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-03-18 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Time to clot engagement | 30 days
  Time from guide catheter placement within the target ICA to clot engagement
Number of device related serious adverse events | Day 1
  Safety profile as measured by number of Intra-procedural device related serious adverse events

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | 90 days post procedure
  0 No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Change in NIH Stroke Scale (NIHSS) | 24 hours
  The score for each ability is a number between 0 (normal functioning) to 4 (completely impaired). The NIHSS has 11 different items and the highest possible score is 42. The higher the score, the more impaired a stroke patient is.
Number of neurovascular guidewires required per case | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Reade De Leacy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No